CLINICAL TRIAL: NCT04925934
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study of VIB7734 for the Treatment of Moderate to Severely Active Systemic Lupus Erythematosus
Brief Title: Study of VIB7734 for the Treatment of Moderate to Severely Active SLE
Acronym: RECAST SLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIB7734.P2.S1; 2020-005528-12 (EudraCT Number)
Record Dates: First submitted 2021-05-04; First posted 2021-06-14 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-arm study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VIB7734 SC (dosing interval 1) (Experimental)
  Interventions: Drug: VIB7734
- VIB7734 SC (dosing interval 2) (Experimental)
  Interventions: Drug: VIB7734
- Placebo SC (dosing interval 3) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VIB7734 — VIB7734
  Other Names: Daxdilimab; HZN-7734
  Arms: VIB7734 SC (dosing interval 1); VIB7734 SC (dosing interval 2)
Other: Placebo — Placebo
  Arms: Placebo SC (dosing interval 3)

SUMMARY:
A Phase 2 Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study of VIB7734 for the Treatment of Moderate to Severely Active Systemic Lupus Erythematosus in approximately 195 participants. The study duration will be 48 weeks, with a safety follow-up through week 56.There will be 3 parallel arms - 2 active treatment and 1 placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years to ≤ 70 years
* Willing and able to understand and provide written informed consent.
* Fulfill the 2019 European League Against Rheumatism/American College of Rheumatology Classification Criteria for SLE
* Disease duration of at least 6 months
* Active SLE as indicated by presence of all the following:

  1. SLEDAI-2K total score ≥ 6 at Screening, excluding fever, SLE headache, or organic brain syndrome.
  2. SLEDAI-2K total score ≥ 4, excluding points attributable to any urine or laboratory results, immunologic measures, fever, SLE headache, or organic brain syndrome at Screening and Baseline (Day 1).
  3. At least one of the following BILAG 2004 Index levels of disease at Screening:
* BILAG A disease in ≥ 1 organ system
* BILAG B disease in ≥ 2 organ systems d. PGA score ≥ 1 on a 0 to 3 visual analog scale (VAS) at Screening

Have at least one of the following at Screening per central lab:

* ANA ≥ 1:80
* Anti-dsDNA antibodies elevated to above normal range as established by the central laboratory (ie, positive results)
* Anti-Smith antibodies elevated to above normal (ie, positive results) Ongoing treatment for SLE

  1. Treatment with one or more disease-modifying anti-rheumatic drug (DMARD) or immunosuppressive medication: Any of the following medications each administered at conventional anti-rheumatic doses for treatment of SLE for at least 12 weeks before Screening (unless discontinued or dose adjusted for documented drug-related toxicity or size/weight), and at a stable dose (including route of administration) for a minimum of 8 weeks prior to Screening and maintained through Baseline (Day 1):
  2. Treatment with OGC monotherapy (without the concomitant use of DMARDs or immunosuppressants):

     * Average daily dose of PO prednisone ≥ 10 mg but ≤ 40 mg (or prednisone equivalent) for a minimum of 4 weeks prior to Screening and a stable dose for minimum of 2 weeks prior to Screening. The dose of OGC must be kept for a minimum of 2 weeks prior to Randomization. Daily dosing or alternate day dosing of PO prednisone or equivalent is allowed.
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at Randomization.
* Non-sterilized male participants who are sexually active with a woman partner of childbearing potential must agree to use a condom with spermicide from Randomization and until 3 months (approximately 5 half-lives) after receipt of the last dose.

Exclusion Criteria:

* Any condition that, in the opinion of the Investigator, or the Sponsor/Central Review Committee, would interfere with the evaluation of the IP or interpretation of participant safety or study results (including borderline disease activity)
* History of allergy, hypersensitivity reaction, or anaphylaxis to any component of the IP or a previous mAb or human Ig therapy
* Active LN or active severe or unstable neuropsychiatric SLE
* Current diagnosis of non-SLE vasculitis syndrome, mixed connective tissue disease, or rheumatic (overlap) syndrome
* Participation in another clinical study with an investigational drug within 4 weeks before Day 1
* Breastfeeding or pregnant women or women who intend to become pregnant anytime from signing the ICF through 6 months after receiving the last dose of IP
* Major surgery within 8 weeks prior to Screening or elective surgery planned from Screening through Day 393.
* Spontaneous or induced abortion, still or live birth, or pregnancy ≤ 4 weeks before Screening
* Known history of a primary immunodeficiency or an underlying condition such as known human immunodeficiency virus (HIV) infection
* Hepatitis B, Hepatitis C, active TB, any severe herpes infection, clinically active infection, or opportunistic infection
* History of clinically significant cardiac disease including unstable angina; and/or myocardial infarction and/or congestive heart failure within 6 months prior to Randomization.
* History of cancer within the past 5 years except, in situ carcinoma of the cervix, cutaneous basal cell or squamous cell carcinoma with curative therapy.
* Receipt of a live-attenuated vaccine within 4 weeks before Day 1 Administration of inactivated (killed) vaccines is acceptable
* The use of immunosuppressants, biologics and DMARDS within the protocol defined washout periods

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen; Nisha Jain, MD, Study Director — Horizon Therapeutics
Locations (67):
- United States (17):
  - Inland Rheumatology Clinical Trials Incorporated, Upland, California
  - Clinical Research of West Florida Inc - Clearwater, Clearwater, Florida
  - Millennium Research, Ormond Beach, Florida
  - IRIS Research and Development LLC, Plantation, Florida
  - Clinical Research of West Florida Inc - Tampa, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Bluegrass Community Research Inc, Lexington, Kentucky
  - NYU Langone Ambulatory Care Brooklyn Heights, Brooklyn, New York
  - Feinstein Institute For Medical Research, Manhasset, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - DJL Clinical Research, Charlotte, North Carolina
  - Paramount Medical Research and Consulting LLC, Middleburg Heights, Ohio
  - Tekton Research Inc, Austin, Texas
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - Spectrum Medical, Inc, Danville, Virginia
- Argentina (7):
  - Consultorios Médicos Dr. Doreski, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Clínica Adventista Belgrano, Estomba, Buenos Aires
  - Framingham Centro Médico, La Plata, Buenos Aires
  - Instituto CER S.A, Quilmes, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes SRL, Quilmes, Buenos Aires
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Consultorio de Investigaciones Reumatologicas, San Miguel de Tucumán, Tucumán Province
- Greece (4):
  - Athens General Hospital 'G Gennimatas, Athens
  - Laiko General Hospital of Athens, Athens
  - University General Hospital of Larissa, Larissa
  - Kianous Stavros, Thessaloniki
- India (5):
  - Krishna Institute of Medical Sciences, Secunderabad, Andhra Pradesh
  - AES - AS - Panchshil Hospital - Ahmedabad, Ahmedabad, Gujarat
  - AES - AS - Unity Trauma Center and ICU - Unity Hospital - Surat, Surat, Gujarat
  - AES - AS - Sushruta Multispeciality Hospital & Research Center Pvt Ltd - Hubli, Hubli, Karnataka
  - Jasleen Hospital, Nagpur, Maharashtra
- Mexico (10):
  - Centro de Investigación en Artritis y Osteoporosis, Mexicali, Estado de Baja California
  - Morales Vargas Centro de Investigacion SC, León, Guanajuato
  - Bioclinica - Centro Integral En Reumatologia Sociedad Anónima de Capital Variable, Guadalajara, Jalisco
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan, Jalisco
  - Centro de Investigación y Tratamiento Reumatológico S.C, San Miguel, Mexico City
  - Centro Peninsular de Investigacion S.C.P, Mérida, Yucatán
  - AMAF Clinical Research,S.C., Distrito Federal
  - Clinica de Investigacion en Reumatologia y Obesidad, Guadalajara
  - Centro de Estudios de Investigacion Basica Y Clinica SC, Jalisco
  - Consultorio de Reumatologia, Mexico City
- Poland (10):
  - Klinika Reumatologii i Rehabilitacji Ortopedyczno-Rehabilitacyjny Szpital Kliniczny im W. Degi, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne Plejady, Krakow, Lesser Poland Voivodeship
  - Pratia MCM, Krakow, Lesser Poland Voivodeship
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól, Lubusz Voivodeship
  - NZOZ Lecznica MAK-MED, Nadarzyn, Masovian Voivodeship
  - Medycyna Kliniczna Marzena Waszczak-Jeka, Warsaw, Masovian Voivodeship
  - Centrum Medyczne AMED, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Czestochowa - PRATIA, Częstochowa, Silesian Voivodeship
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz
  - Centrym Medyczne AMED oddzial w Lodzi, Lodz, Łódź Voivodeship
- Russia (3):
  - Belyayev Clinical Hospital of the Kuzbass, Kemerovo
  - O.M. Filatov City Clinical Hospital #15, Moscow
  - Departmental Hospital at Smolensk Station "rzhd" JSC, Smolensk
- Serbia (3):
  - Institute of Rheumatology Belgrade, Belgrade
  - Military Medical Academy, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
- Spain (2):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Quironsalud Infanta Luisa, Seville
- Taiwan (3):
  - Kaohsiung Veterans General Hospital, Kaohsiung City, Province of China
  - National Taiwan University Hospital, Taipei, Province of China
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District, Province of China
- Ukraine (3):
  - Medical Center of LLC Modern Clinic, Zaporizhzhia, Zaporizhzhia Oblast
  - Limited Liability Company Medical Center Consilium, Kiyiv
  - ME Poltava Reg.Clin.Hospital n.a.M.V.Skliphosovskyi of Poltava Reg.Council, Poltava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with systemic lupus erythematosus (SLE) were enrolled at 68 sites in the United States, Argentina, Greece, India, Mexico, Poland, Serbia, Spain, Taiwan, Ukraine and Russia between May 2021 and June 2023.
Pre-assignment Details: Participants were randomized in a 1:1:1 ratio to take daxdilimab 200 mg every 4 weeks (Q4W) subcutaneously (SC), daxdilimab 200 mg every 12 weeks (Q12W) SC (with an additional 200 mg SC dose at Week 4) or matching placebo Q4W SC. Duration of treatment was up to 48 weeks. Randomization was stratified by SLE Disease Activity Index 2000 (SLEDAI-2K) total score at screening (≥ 10 or < 10) and prednisone or equivalent oral glucocorticoid (OGC) dose at baseline (≥ 10 mg/day or < 10 mg/day).
Groups:
- Placebo: Participants were randomized to receive matching placebo Q4W SC for a treatment period up to 48 weeks.
- Daxdilimab 200 mg Q4W: Participants were randomized to receive daxdilimab 200 mg Q4W for a treatment period up to 48 weeks.
- Daxdilimab 200 mg Q12W: Participants were randomized to receive daxdilimab 200 mg Q12W (with an additional 200 mg SC dose at Week 4) for a treatment period up to 48 weeks.
Period: Overall Study
Arm/Group | Placebo | Daxdilimab 200 mg Q4W | Daxdilimab 200 mg Q12W
Started | 71 | 72 | 71
Completed | 51 | 61 | 57
Not Completed | 20 | 11 | 14
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Withdrawal by Subject | 8 | 5 | 9
Not completed — Other | 2 | 2 | 2
Not completed — Eastern European Conflict | 7 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): included all randomized participants who received any dose of investigational product (IP). Participants were analyzed according to the treatment randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Daxdilimab 200 mg Q4W | Daxdilimab 200 mg Q12W | Total
Number analyzed (Participants) | 71 | 72 | 71 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (11.0) | 44.5 (13.1) | 45.3 (11.6) | 43.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 67 | 66 | 200
  Male | 4 | 5 | 5 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 2 | 2 | 0 | 4
  Asian | 9 | 7 | 10 | 26
  Black or African American | 4 | 8 | 6 | 18
  White | 54 | 49 | 51 | 154
  Other | 1 | 6 | 4 | 11
  Multiple categories checked | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 25 | 27 | 27 | 79
  Not Hispanic or Latino | 46 | 45 | 44 | 135
Number of Participants Within Each OGC Stratification Dose Level [Number; unit: number of participants] — OGC dose represents the baseline dose of prednisone or any equivalent corticosteroids.
  number of participants
    < 10 mg/day | 36 | 35 | 36 | 107
    ≥ 10 mg/day | 35 | 37 | 35 | 107
SLEDAI-2K Score [Mean (Standard Deviation); unit: Score] — The SLEDAI-2K assessment consists of 24 lupus-related items. It is a weighted instrument, in which descriptors are multiplied by an organ's "weight". For example, renal descriptors are multiplied by 4 and CNS descriptors by 8; these weighted organ manifestations are totalled into the final score. The scores range from 0 to 105, with higher scores indicating more severe disease activity.
  Score | 9.9 (2.8) | 10.6 (4.0) | 10.1 (2.9) | 10.2 (3.3)
British Isles Lupus Assessment Group (BILAG)-2004 Score [Mean (Standard Deviation); unit: scores on a scale] — The BILAG-2004 Index assesses lupus disease activity across 9 organ systems. Each organ system is graded from A (severe disease activity requiring urgent treatment; score of 12) to E (system never involved; score of 0). The organ system scores are summed to give an overall score ranging from 0 to 108 where higher scores indicate greater disease activity and severity.
  scores on a scale | 19.2 (4.7) | 19.5 (4.6) | 19.8 (5.5) | 19.5 (4.9)
Physician Global Assessment (PGA) Score [Median (Standard Deviation); unit: Score] — The PGA takes into account various clinical factors, including the participant's symptoms, physical examination findings, laboratory results, and the physician's judgment. The PGA is scored with a range 0 to 3 where higher scores indicate greater disease activity and severity.
  Score | 1.89 (0.37) | 1.96 (0.32) | 1.90 (0.41) | 1.91 (0.37)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving a BILAG-2004 Index-based Combined Lupus Assessment (BICLA) Response and an OGC Dose ≤ 7.5 mg/Day and ≤ Baseline Dose of Prednisone or Equivalent at Week 48
Description: A BICLA response required improvement in all domains affected at baseline, assessed by the BILAG 2004, no worsening of other BILAG 2004 domains, no worsening of SLEDAI-2K or PGA scores compared with baseline, no use of restricted medications beyond the protocol-allowed threshold, and no discontinuation of IP.
Time Frame: Week 48
Population: FAS: included all randomized participants who received any dose of IP. Participants were analyzed according to the treatment randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Daxdilimab 200 mg Q4W | Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 64 | 69 | 69
Participants | 25 | 29 | 27
Statistical Analysis 1: Comparison: Placebo vs Daxdilimab 200 mg Q4W; Adjusted response rate, rate difference and p-value are from logistic regression analysis with treatment and randomization stratification factors in the model; Test type: Superiority; p = 0.7474, Regression, Logistic; Rate Difference = 2.8, 90% CI 2-sided [-11.4 to 17.0]
Statistical Analysis 2: Comparison: Placebo vs Daxdilimab 200 mg Q12W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9942, Regression, Logistic; Rate Difference = -0.1, 90% CI 2-sided [-14.2 to 14.1]

2. Secondary Outcome: Number of Participants With a Cutaneous Lupus Erythematosus Disease Area and Severity Index-Activity (CLASI-A) Score ≥ 10 at Baseline Achieving ≥ 50% Reduction From Baseline in CLASI-A Score at Week 12
Description: The CLASI-A evaluates erythema (0-3 [higher scores indicate more severe redness]), scale/hypertrophy (0-2 [higher scores indicate more extensive scaling/thickening]), mucous membrane lesions (0 [absent] or 1 [present]), recent hair loss (0 [absent] or 1 [present]), and non-scarring alopecia (0-3 [(higher scores indicate more extensive hair loss without scarring]) at 13 anatomical sites on the skin. Total score is calculated by summing scores across all anatomical locations for each parameter. Higher total scores indicate greater disease activity and severity in SLE. Reduction of 50% in CLASI-A score was defined by meeting all the following conditions:
  1. A ≥ 50% reduction of CLASI-A score at Week 12 as compared to baseline.
  2. No use of restricted medications beyond the protocol-allowed threshold before assessment.
  3. No discontinuation of IP.
Time Frame: Week 12
Population: FAS: included all randomized participants who received any dose of IP. Participants were analyzed according to the treatment randomized. Only participants with a CLASI-A score ≥ 10 at baseline were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Daxdilimab 200 mg Q4W | Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 8 | 10 | 14
Participants | 1 | 4 | 5
Statistical Analysis 1: Comparison: Placebo vs Daxdilimab 200 mg Q4W; Adjusted response rate, rate difference and p-value are from logistic regression analysis with treatment, randomization stratification factors and Baseline CLASI-A score in the model; Test type: Superiority; p = 0.1626, Regression, Logistic; Rate Difference = 37.2, 90% CI 2-sided [-0.3 to 74.7]
Statistical Analysis 2: Comparison: Placebo vs Daxdilimab 200 mg Q12W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2873, Regression, Logistic; Rate Difference = 24.1, 90% CI 2-sided [-7.5 to 55.8]

3. Secondary Outcome: Number of Participants Achieving an SLE Responder Index (SRI)-4 Response and an OGC Dose ≤ 7.5 mg/Day and ≤ Baseline Dose of Prednisone or Equivalent at Week 48
Description: The SRI-4 measures reduction in SLE disease activity and it is a composite measure that includes the SLEDAI-2K, BILAG-2004, and PGA. SRI responder was defined by meeting all of the following criteria: 1) Reduction of ≥4 points from baseline in SLEDAI-2K score; 2) no new BILAG A or no more than 1 new BILAG B disease activity scores and 3) no worsening (defined as an increase of ≥0.3 points [0-3 scale] from baseline) in the PGA.
Time Frame: Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Daxdilimab 200 mg Q4W | Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 64 | 69 | 69
Participants | 26 | 34 | 30
Statistical Analysis 1: Comparison: Placebo vs Daxdilimab 200 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3220, Regression, Logistic; Rate Difference = 8.6, 90% CI 2-sided [-5.6 to 22.7]
Statistical Analysis 2: Comparison: Placebo vs Daxdilimab 200 mg Q12W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7364, Regression, Logistic; Rate Difference = 2.9, 90% CI 2-sided [-11.2 to 17.0]

4. Secondary Outcome: Number of Participants With an OGC Dose ≥ 10 mg/Day of Prednisone or Equivalent at Baseline Who Maintained an OGC Dose ≤ 7.5 mg/Day From Week 36 Through Week 48
Description: Maintenance of OGC reduction from Week 36 to Week 48 was defined by meeting all the following criteria:
  1. Achieved an OGC dose of ≤ 7.5 mg/day prednisone or equivalent at Week 36
  2. Maintained an OGC dose of ≤ 7.5 mg/day from Week 36 through Week 48
  3. No use of restricted medications beyond the protocol-allowed threshold before assessment
  4. No discontinuation of IP before assessment
Time Frame: Week 36 up to Week 48
Population: FAS: included all randomized participants who received any dose of IP. Participants were analyzed according to the treatment randomized. Data excludes participants from Russia and Ukraine sites. Only participants with an OGC dose ≥ 10 mg/day of prednisone or equivalent at baseline were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Daxdilimab 200 mg Q4W | Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 30 | 34 | 34
Participants | 20 | 27 | 26
Statistical Analysis 1: Comparison: Placebo vs Daxdilimab 200 mg Q4W; Adjusted response rate, rate difference and p-value are from logistic regression analysis with treatment, stratification factors (SLEDAI-2K only) and Baseline OGC dose included in the model; Test type: Superiority; p = 0.2805, Regression, Logistic; Rate Difference = 11.7, 90% CI 2-sided [-6.1 to 29.4]
Statistical Analysis 2: Comparison: Placebo vs Daxdilimab 200 mg Q12W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.3926, Regression, Logistic; Rate Difference = 9.4, 90% CI 2-sided [-8.6 to 27.3]

5. Secondary Outcome: Number of Participants Achieving Lupus Low Disease Activity State (LLDAS) at Week 48
Description: LLDAS was defined by meeting all of the following criteria:
  1. SLEDAI-2K ≤ 4, with no activity in major organ systems (renal, central nervous system, cardiopulmonary, vasculitis, fever) and no hemolytic anemia or gastrointestinal activity measured as maintaining a D (no disease activity but suggests the system had previously been affected) or E (no current or previous disease activity) score in BILAG Gastrointestinal Body System
  2. No new lupus disease activity compared with the previous
  3. Physician's Global Assessment of Disease Activity ≤ 1 on a 3-point visual analog scale from no disease activity to severe disease activity
  4. A current prednisolone (or equivalent) dose ≤ 7.5 mg daily
  5. Well-tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents
Time Frame: Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Daxdilimab 200 mg Q4W | Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 64 | 69 | 69
Participants | 11 | 23 | 15
Statistical Analysis 1: Comparison: Placebo vs Daxdilimab 200 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0370, Regression, Logistic; Rate Difference = 16.5, 90% CI 2-sided [4.0 to 29.0]
Statistical Analysis 2: Comparison: Placebo vs Daxdilimab 200 mg Q12W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4939, Regression, Logistic; Rate Difference = 4.9, 90% CI 2-sided [-6.7 to 16.4]

6. Secondary Outcome: Serum Concentration of Daxdilimab
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48
Population: Pharmacokinetic (PK) analysis set: included all participants who received any dose of daxdilimab in the study and had at least 1 quantifiable serum PK observation post-first dose. Participants were analyzed according to the treatment that they received.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Placebo | Daxdilimab 200 mg Q4W | Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 0 | 72 | 71
ug/mL
  Baseline |  | 0.011 (0.026) | 0.008 (0.004)
  Week 4: number analyzed (Participants) | 0 | 71 | 71
  Week 4 |  | 3.319 (1.972) | 3.301 (1.718)
  Week 8 |  | 4.714 (3.079) | 4.643 (2.708)
  Week 12: number analyzed (Participants) | 0 | 70 | 70
  Week 12 |  | 5.344 (3.624) | 1.372 (1.189)
  Week 16: number analyzed (Participants) | 0 | 68 | 65
  Week 16 |  | 5.035 (3.377) | 4.268 (2.720)
  Week 20: number analyzed (Participants) | 0 | 66 | 64
  Week 20 |  | 5.884 (4.451) | 1.239 (1.097)
  Week 24: number analyzed (Participants) | 0 | 63 | 62
  Week 24 |  | 5.539 (4.224) | 0.530 (0.922)
  Week 28: number analyzed (Participants) | 0 | 65 | 61
  Week 28 |  | 4.855 (3.743) | 3.590 (2.522)
  Week 32: number analyzed (Participants) | 0 | 65 | 61
  Week 32 |  | 4.951 (4.047) | 1.096 (1.151)
  Week 36: number analyzed (Participants) | 0 | 63 | 59
  Week 36 |  | 5.321 (4.309) | 0.366 (0.471)
  Week 40: number analyzed (Participants) | 0 | 65 | 59
  Week 40 |  | 4.652 (3.426) | 3.439 (2.534)
  Week 44: number analyzed (Participants) | 0 | 64 | 59
  Week 44 |  | 4.908 (3.780) | 1.115 (1.378)
  Week 48: number analyzed (Participants) | 0 | 60 | 58
  Week 48 |  | 5.543 (4.637) | 0.406 (0.585)

7. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) to Daxdilimab
Description: A baseline ADA-positive participant was defined as a participant who had an ADA positive sample at baseline. ADA incidence is the number of the participants ADA positive post-Baseline only or who boosted their preexisting ADA (≥ 4 × Baseline level) during the trial. Persistent positive was defined as ADA positive at ≥ 2 post-Baseline assessments (with ≥ 16 weeks between first and last positive) or positive at last post-Baseline assessment. Transient positive was defined as ADA post-Baseline positive but did not fulfill the criteria of persistent positive.
Time Frame: Baseline to Week 56
Population: Safety analysis set (SAS): included all participants who received any dose of IP. Participants were analyzed according to the treatment that they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Daxdilimab 200 mg Q4W | Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 71 | 72 | 71
Participants
  ADA not detected (negative) on trial | 47 | 59 | 56
  ADA incidence | 14 | 6 | 6
  Boosted ADA (≥ 4 × Baseline level) | 1 | 2 | 2
  ADA detected (positive) on trial: ADA prevalence | 24 | 13 | 15
  Only Baseline positive | 1 | 5 | 5
  Only post-Baseline positive | 13 | 4 | 4
  Both Baseline and post-Baseline positive | 10 | 4 | 6
  Persistent positive | 19 | 8 | 8
  Transient positive | 4 | 0 | 2

8. Secondary Outcome: Change From Baseline in Plasmacytoid Dendritic Cell (pDCs) Expression in Blood
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 20, Week 24, Week 32, Week 36, Week 44, Week 48, Week 52, Week 56
Population: SAS: included all participants who received any dose of IP. Participants were analyzed according to the treatment that they received. Only participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Placebo | Daxdilimab 200 mg Q4W | Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 43 | 48 | 46
cells/uL
  Baseline | 2.5068 (1.8486) | 2.2960 (1.7457) | 1.9195 (1.1990)
  Week 4: number analyzed (Participants) | 33 | 42 | 41
  Week 4 | -0.2324 (1.8194) | -1.4240 (1.9493) | -1.2903 (1.2201)
  Week 8: number analyzed (Participants) | 32 | 43 | 38
  Week 8 | -0.4608 (1.4125) | -1.5194 (1.7555) | -1.1486 (1.2090)
  Week 12: number analyzed (Participants) | 33 | 42 | 39
  Week 12 | 0.0275 (1.7580) | -1.5164 (1.8180) | -1.1134 (1.5290)
  Week 20: number analyzed (Participants) | 32 | 43 | 35
  Week 20 | 285.1519 (1613.566) | -1.5131 (1.6837) | -1.0320 (1.1063)
  Week 24: number analyzed (Participants) | 30 | 40 | 40
  Week 24 | -0.3911 (1.7344) | -1.5974 (1.7705) | -0.5507 (1.3090)
  Week 32: number analyzed (Participants) | 26 | 40 | 38
  Week 32 | 0.3513 (1.7855) | -1.3367 (1.5678) | -0.8496 (1.2403)
  Week 36: number analyzed (Participants) | 26 | 37 | 33
  Week 36 | -0.1274 (1.6962) | -1.4614 (1.7634) | -0.9131 (0.9845)
  Week 44: number analyzed (Participants) | 28 | 39 | 33
  Week 44 | -0.3194 (1.6347) | -1.6540 (1.6184) | -1.1322 (1.3782)
  Week 48: number analyzed (Participants) | 28 | 36 | 36
  Week 48 | 0.1973 (2.4112) | -1.4608 (1.5647) | -0.7964 (1.0055)
  Week 52: number analyzed (Participants) | 3 | 3 | 7
  Week 52 | 0.1483 (3.7955) | -0.4353 (0.5127) | 0.0149 (0.7999)
  Week 56: number analyzed (Participants) | 3 | 3 | 5
  Week 56 | -2.0823 (3.9807) | -2.3137 (3.2514) | -0.7056 (0.6729)

9. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of an intervention in humans whether or not it is considered intervention-related. TEAEs are AEs that started on or after the first dose of IP. An AE was considered serious (SAE) if it resulted in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolonged existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, a congenital abnormality/birth defect, or an important medical event. AE severity was rated according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0: grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (life-threatening), grade 5 (death).
Time Frame: Up to Week 56
Population: SAS: included all participants who received any dose of IP. Participants were analyzed according to the treatment that they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Daxdilimab 200 mg Q4W | Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 71 | 72 | 71
Participants
  TEAEs | 49 | 49 | 58
  Treatment-related TEAEs | 10 | 17 | 17
  AEs Grade 3 or higher | 5 | 8 | 9
  SAEs | 8 | 9 | 9
  Treatment-related SAEs | 0 | 1 | 0
  AEs Resulting in Death | 0 | 1 | 0

10. Secondary Outcome: Number of Participants Who Experienced AEs of Special Interest (AESI)
Description: An AESI is an AE of scientific and medical interest specific to understanding of the IP and may require close monitoring and collection of additional information by the Investigator. AESIs for this study included:
  1. Hypersensitivity reaction, including anaphylaxis.
  2. Severe (Grade 3 or higher) viral infections/reactivations.
  3. Opportunistic infection.
  4. Malignancy (except non-melanoma skin cancer).
Time Frame: Up to Week 56
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Daxdilimab 200 mg Q4W | Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 71 | 72 | 71
Participants
  Hypersensitivity Reaction Including Anaphylaxis | 1 | 0 | 1
  Opportunistic infection | 1 | 1 | 1
  Viral infection/Reactivation | 10 | 6 | 7

ADVERSE EVENTS:
Time Frame: Up to 56 weeks
Description: SAS: included all participants who received any dose of IP. Participants were analyzed according to the treatment that they received. All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Daxdilimab 200mg Q4W: Participants were randomized to receive daxdilimab 200 mg Q4W for a treatment period up to 48 weeks.
- Daxdilimab 200mg Q12W: Participants were randomized to receive daxdilimab 200 mg Q12W (with an additional 200 mg SC dose at Week 4) for a treatment period up to 48 weeks.
Arm/Group | Placebo | Daxdilimab 200mg Q4W | Daxdilimab 200mg Q12W
All-Cause Mortality (participants affected / at risk) | 0/71 | 1/72 | 0/71
Serious Adverse Events (participants affected / at risk) | 8/71 | 9/72 | 9/71
Other Adverse Events (participants affected / at risk) | 17/71 | 30/72 | 29/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | Daxdilimab 200mg Q4W (N=72) | Daxdilimab 200mg Q12W (N=71)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Huntington's disease (Congenital, familial and genetic disorders) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Abortion induced incomplete (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Hydrosalpinx (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | Daxdilimab 200mg Q4W (N=72) | Daxdilimab 200mg Q12W (N=71)
Palpitations (Cardiac disorders) | 0 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 4
COVID-19 (Infections and infestations) | 9 | 10 | 9
Influenza (Infections and infestations) | 0 | 4 | 2
Nasopharyngitis (Infections and infestations) | 4 | 3 | 2
Sinusitis (Infections and infestations) | 1 | 4 | 2
Upper respiratory tract infection bacterial (Infections and infestations) | 2 | 1 | 4
Urinary tract infection (Infections and infestations) | 4 | 7 | 8
Headache (Nervous system disorders) | 5 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT04925934/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT04925934/SAP_001.pdf